CLINICAL TRIAL: NCT01432327
Title: The Impact of Real-time Feedback on Physical Activity Patterns in Flemish Employees: an Intervention Study
Brief Title: The Impact of Real-time Feedback on Physical Activity Patterns in Flemish Employees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Karen Van Hoye, Phd Student, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KULEUVEN_RTFDB
Record Dates: First submitted 2011-09-09; First posted 2011-09-12 (Estimated); Results first posted 2012-04-18 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-02

CONDITIONS: Sedentary Lifestyle
Keywords: motor activity; randomized controlled trial; feedback
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control group (Placebo Comparator): This group receives no kind of feedback during the intervention period. The participants wear the SenseWear Armband for 4 weeks and results of the intervention are discussed after the 4 week intervention period.
  Interventions: Device: SenseWear Armband
- Step Group (Experimental): This group receives feedback about the daily amount of steps by means of a pedometer.
  Interventions: Device: Pedometer
- Display Group (Experimental): Participants receive real time feedback on their energy expenditure, minutes of physical activity and step count by means of the SenseWear Display
  Interventions: Device: SenseWear display
- Coaching Group (Experimental): Participants receive real-time feedback on their energy expenditure, step count and minutes of physical activity by means of the SenseWear Display and weekly meet with a Personal Coach to discuss their progress
  Interventions: Behavioral: Personal Coaching

INTERVENTIONS:
Device: SenseWear display — Participants use the self-monitoring device (display) to aid behavior change via real-time lifestyle feedback targeting physical activity.
  The display has a versatile design that allows it to be clipped to a shirt, bag or belt loop. The Display can help participants stay in sync with their daily goals.
  Other Names: BodyMedia® Display (Model DD100)
  Arms: Display Group
Device: Pedometer — Participants receive a pedometer to determine their daily amount of steps. Every day they write down their amount of steps in a step diary.
  Other Names: Yamax Digi-Walker SW-200
  Arms: Step Group
Device: SenseWear Armband — Participants wear the SenseWear Armband for 4 weeks
  Other Names: SenseWear Pro3 Armband; BodyMedia, Inc. Pittsburgh, PA
  Arms: Control group
Behavioral: Personal Coaching — A weekly meeting with a Personal Coach to evaluate the physical activity patterns in daily life
  Arms: Coaching Group

SUMMARY:
The aim of the study is to assess an increase of daily physical activity from electronic self-monitoring, to compare these values to the 10.000 step program, and to compare with real-time feedback with and without guidance from a Personal Coach.

DETAILED DESCRIPTION:
The purpose of this intervention study is to determine the effectiveness of continuous self-monitoring and real-time feedback from the SenseWear Armband (BodyMedia) alone and in combination with Personal Coaching to enhance physical activity and influence consciousness about its own physical activity patterns over a 12-month period in sedentary Flemish employees. The investigators hypothesize that the use of the feedback will increase awareness and subsequent physical activity levels of inactive office workers. Another hypothesizes is that the weekly meeting with a Personal Coach will add a controlling element and therefore employees of the 'coaching group' will have a higher physical activity level at the end of the intervention period compared to the other groups.

ELIGIBILITY:
Inclusion Criteria:

* Employee
* Physical Activity Level < 1.71 MET
* Willing to wear the SenseWear Armband for 5-6 weeks

Exclusion Criteria:

* Student
* Senior

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2010-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johan Lefevre, Prof Dr., Study Director — KU Leuven
Locations (1):
- Katholieke Universiteit Leuven - Tervuursevest 101, Leuven, Belgium

REFERENCES:
- [Derived] Van Hoye K, Wijtzes AI, Lefevre J, De Baere S, Boen F. Year-round effects of a four-week randomized controlled trial using different types of feedback on employees' physical activity. BMC Public Health. 2018 Apr 12;18(1):492. doi: 10.1186/s12889-018-5402-0. PMID 29649997

RESULTS

PARTICIPANT FLOW:
Recruitment Details: August 2010 - May 2010: recruitement of employees. Method: flyering at Pharmacists, word of mouth, information session at companies in and around the region of Antwerp
Pre-assignment Details: Students and seniors were excluded from the study. Participants with an average Physical Activity Level above 1.71 times their resting metabolic rate were excluded from the trial
Groups:
- Control Group: This group receives no kind of feedback during the intervention period
Period: Baseline
Arm/Group | Control Group | Step Group | Display Group | Coaching Group
Started | 56 | 57 | 57 | 57
Completed | 56 | 57 | 57 | 57
Not Completed | 0 | 0 | 0 | 0
Period: Posttest 3 Months
Arm/Group | Control Group | Step Group | Display Group | Coaching Group
Started | 56 | 57 | 57 | 57
Completed | 52 | 55 | 55 | 56
Not Completed | 4 | 2 | 2 | 1
Not completed — depression | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2 | 1
Not completed — Allergic reaction | 0 | 2 | 0 | 0
Period: Posttest 6 Months
Arm/Group | Control Group | Step Group | Display Group | Coaching Group
Started | 52 | 55 | 55 | 56
Completed | 52 | 55 | 50 | 54
Not Completed | 0 | 0 | 5 | 2
Not completed — Lost to Follow-up | 0 | 0 | 3 | 2
Not completed — Allergic reaction | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: Posttest 1 Year
Arm/Group | Control Group | Step Group | Display Group | Coaching Group
Started | 52 | 55 | 50 | 54
Completed | 28 | 27 | 30 | 31
Not Completed | 24 | 28 | 20 | 23
Not completed — Measurement have to take place in future | 24 | 28 | 15 | 20
Not completed — Lost to Follow-up | 0 | 0 | 4 | 2
Not completed — Allergic reaction | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Step Group | Display Group | Coaching Group | Total
Number analyzed (Participants) | 56 | 57 | 57 | 57 | 227
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 56 | 57 | 57 | 57 | 227
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (11) | 43 (11) | 44 (10) | 41 (10) | 41 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 31 | 31 | 124
  Male | 25 | 26 | 26 | 26 | 103
Region of Enrollment [Number; unit: participants]
  Belgium | 56 | 57 | 57 | 57 | 227

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity Level
Description: To account for differences in body size and composition, the 24-hour energy requirement (kcal/day) is expressed as a multiple of the basal metabolic rate per 24 hours by using the PAL value (PAL = total energy expenditure/basal metabolic rate). A desirable PAL includes the regular practice of physical activity at work or in spare time with an intensity and duration that will reduce the risk of becoming overweight and developing a variety of non-communicable chronic diseases usually associated as co-morbidities with obesity. This corresponds to PAL values of 1.75 and higher.
Time Frame: One year
Population: Intention to treat analysis was used and analyses data from all participants, including those who did not complete the study
Measure: Mean (Standard Deviation); unit: Metabolic Equivalent
Arm/Group | Control Group | Step Group | Display Group | Coaching Group
Number analyzed (Participants) | 55 | 56 | 57 | 56
Metabolic Equivalent | 1.45 (0.15) | 1.40 (0.16) | 1.46 (0.17) | 1.46 (0.18)

2. Secondary Outcome: Daily Energy Expenditure in Physical Activity
Description: Minutes of physical activity. Activities can be classified as moderate-intensity, vigorous-intensity or very vigorous-intensity activities based upon the amount of energy used by the body while doing the activity.
Time Frame: One year
Reporting Status: Not Posted

3. Secondary Outcome: Percent of Participants Losing Fat Percentage
Description: The amount of body fat is measured by bioelectrical impedance analysis (BIA).
Time Frame: One Year
Reporting Status: Not Posted

4. Secondary Outcome: Stages of Motivational Readiness for Physical Activity
Description: According to The Stages of Motivational Readiness for Change Model (SOC), individuals move through a series of stages as they adopt and maintain a new habit(Prochaska & DiClemente, 1983). Specifically, the stages include Precontemplation, Contemplation, Preparation, Action, and Maintenance.The relevant variables were assessed in a self-administered questionnaire.
Time Frame: One Year
Reporting Status: Not Posted

5. Secondary Outcome: Step Count
Description: Daily number of steps
Time Frame: One Year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Participants were followed for a time period of 1 year.
Description: The risk of an adverse cardiovascular event occurring during or following an acute bout of PA is greatest among new exercisers who are formerly sedentary and/or who display certain disease risk factors. The intervention did not result in any observable occurrences that has unfavorable and/or unintended effects on research subjects.
Arm/Group | Control Group | Step Group | Display Group | Coaching Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 0/56 | 0/57 | 0/57 | 0/57

LIMITATIONS AND CAVEATS:
Malfunction of the SenseWear Armband: 4 out of the 320 baseline measurements

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No